CLINICAL TRIAL: NCT00266409
Title: A Multicenter, Randomized, Open-label, Parallel Design Trial to Compare Time to Response in the Symptoms of Anxiety to Concomitant Treatment With Niravam™ and an SSRI or SNRI to Treatment With an SSRI or SNRI Alone in Subjects With Generalized Anxiety Disorder or Panic Disorder
Brief Title: Trial to Compare Time to Response in the Symptoms of Anxiety to Concomitant Treatment With Niravam™ and an SSRI or SNRI to Treatment With an SSRI or SNRI Alone in Subjects With Generalized Anxiety Disorder or Panic Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SP0851
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Results first posted 2009-10-02 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2009-12

CONDITIONS: Generalized Anxiety Disorder; Panic Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder; Panic Disorder | interventions — Alprazolam

ARMS (4):
- Panic: Niravam+SSRI/SNRI (Experimental): Panic Disorder: Niravam plus a newly prescribed SSRI or SNRI
  Interventions: Drug: Niravam; Drug: SSRI/SNRI
- Panic: SSRI/SNRI alone (Experimental): Panic Disorder: Newly prescribed SSRI or SNRI alone
  Interventions: Drug: SSRI/SNRI
- GAD: Niravam+SSRI/SNRI (Experimental): Generalized Anxiety Disorder: Niravam plus a newly prescribed SSRI or SNRI
  Interventions: Drug: Niravam; Drug: SSRI/SNRI
- GAD: SSRI/SNRI alone (Experimental): Generalized Anxiety Disorder: Newly prescribed SSRI or SNRI alone
  Interventions: Drug: SSRI/SNRI

INTERVENTIONS:
Drug: Niravam
  Other Names: Alprazolam
  Arms: GAD: Niravam+SSRI/SNRI; Panic: Niravam+SSRI/SNRI
Drug: SSRI/SNRI — Selective Serotonin Reuptake Inhibitor or Selective Norepinephrine Reuptake Inhibitor

SUMMARY:
An 8-week, open-label trial in 848 subjects at 212 sites to compare time to response in symptoms of anxiety in subjects treated with Niravam™ and a newly prescribed Selective Serotonin Reuptake Inhibitor (SSRI)or Serotonin and Norepinephrine Reuptake Inhibitor (SNRI) to that in subjects treated with a newly prescribed SSRI/SNRI alone. Subjects must be at least 18 years of age and positive for Generalized Anxiety Disorder (GAD)or Panic Disorder. Subjects will be randomized to receive concomitant Niravam™ and an SSRI/SNRI or an SSRI/SNRI alone during the study. Most symptom evaluations will be done using an automated phone interview system. There are 4 clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age.
* Diagnosed by the Investigator with primary Generalized Anxiety Disorder (GAD) and/or primary Panic Disorder with or without agoraphobia, either primary episode or recurrence, and is positive for GAD or Panic Disorder by the MHS (Mental Health Screener)).
* Receiving a new prescription for all SSRI or SNRI as indicated for GAD or Panic Disorder with or without agoraphobia. Definition of a new prescription in case of a recurrence in symptoms is no prescription or refill of prescription of SSRI or SNRI for the past 6 months.
* Subject is informed and given ample time and opportunity to think about his/her participation and has given his/her written informed consent.

Exclusion Criteria:

* Presence of medical condition or presence of schizophrenia, bipolar disorder, alcohol abuse/dependence or any other primary major psychiatric disorder that, in the opinion of the Investigator, would jeopardize the subject or compromise the subject's ability to participate in the trial.
* Is a current suicide risk in the opinion of the Investigator.
* Has initiated cognitive therapy within two months of Study Day 1.
* Does not speak English or does not hear well enough to be able to perform the Hamilton Anxiety (HAM-A) Rating Scale and Mental Health Screener (MHS) by Interactive Voice Response System (IVRS).
* Has taken a benzodiazepine within the past 30 days.
* History of hypersensitivity or allergic response to any of the components of SSRIs, SNRIs, benzodiazepines, or related drugs.
* If a female of child-bearing potential, is pregnant, nursing, or not using appropriate birth control methods.
* Presence of contraindications to the SSRI or SNRI to be prescribed per the specific package insert.
* Presence of acute narrow angle glaucoma or taking ketoconazole or itraconazole,which are contraindications to Niravam per the package insert.
* History of phenylketonuria (PKU).
* Participation in a previous clinical trial within 30 days prior to Study Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2005-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (1):
- Schwarz, Milwaukee, Wisconsin, United States

REFERENCES:
- [Result] Katzelnick DJ, Saidi J, Vanelli MR, Jefferson JW, Harper JM, McCrary KE. Time to response in panic disorder in a naturalistic setting: combination therapy with alprazolam orally disintegrating tablets and serotonin reuptake inhibitors compared to serotonin reuptake inhibitors alone. Psychiatry (Edgmont). 2006 Dec;3(12):39-49. PMID 20877555
- [Result] Rapaport MH, Skarky SB, Katzelnick DJ, Dewester JN, Harper JM, McCrary KE. Time to response in generalized anxiety disorder in a naturalistic setting: combination therapy with alprazolam orally disintegrating tablets and serotonin reuptake inhibitors compared to serotonin reuptake inhibitors alone. Psychiatry (Edgmont). 2006 Dec;3(12):50-9. PMID 20877556
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants Flow shows 418 subjects that have been enrolled and randomized. The safety population consists of 414 subjects that received at least one dose of SSRI/SNRI and/or Niravam.
Pre-assignment Details: Baseline Characteristics are only available for the Intent-to-treat population (subjects who received one dose of SSRI/SNRI and/or Niravam and have an assessment beyond the Baseline assessment)
Groups:
- GAD : Niravam+SSRI/SNRI: Generalized Anxiety Disorder: Niravam plus newly prescribed SSRI or SNRI
Period: Overall Study
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Started | 137 | 138 | 72 | 71
Completed | 92 | 92 | 55 | 49
Not Completed | 45 | 46 | 17 | 22
Not completed — Lack of Efficacy | 2 | 6 | 1 | 2
Not completed — Adverse Event | 7 | 2 | 1 | 1
Not completed — Lost to Follow-up | 18 | 21 | 6 | 8
Not completed — Withdrawal by Subject | 6 | 10 | 3 | 9
Not completed — Protocol Violation | 5 | 3 | 4 | 2
Not completed — Other | 7 | 4 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone | Total
Number analyzed (Participants) | 125 | 120 | 67 | 62 | 374
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 120 | 119 | 66 | 61 | 366
  >=65 years | 5 | 1 | 1 | 1 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (12.24) | 38.1 (12.55) | 40.1 (12.64) | 43.6 (12.20) | 40 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 93 | 50 | 42 | 287
  Male | 23 | 27 | 17 | 20 | 87
Region of Enrollment [Number; unit: participants]
  United States | 125 | 120 | 67 | 62 | 374

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Percent of Participants Showing a Response in the Symptoms of Anxiety (Decrease in Total Hamilton Anxiety (HAM-A) -Score of >=50%) in the Intent-to-treat Population (Kaplan-Meier-estimates)
Description: The Hamilton Anxiety (HAM-A) Rating scale is a test of 14 items measuring the severity of anxiety symptoms. Each item is rated on a 5-point ordinal scale, ranging from 0 (not present) to 4 (severe). Thus total possible score is 56. Kaplan-Meier-analysis was performed and Kaplan-Meier estimates (cumulative percent of subjects responding) are presented.
Time Frame: 10 weeks
Population: Intent-to-treat population
Measure: Number; unit: cumulative percent of responders
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 125 | 120 | 67 | 62
cumulative percent of responders
  Week 1 | 1.60 | 0.83 | 1.49 | 1.61
  Week 2 | 3.20 | 21.73 | 32.93 | 27.52
  Week 3 | 45.83 | 39.43 | 51.22 | 48.89
  Week 4 | 59.22 | 52.40 | 57.32 | 62.14
  Week 5 | 69.68 | 65.99 | 66.47 | 65.92
  Week 6 | 71.57 | 69.79 | 69.66 | 71.94
  Week 7 | 74.59 | 74.11 | 74.66 | 73.94
  Week 8 | 76.62 | 76.27 | 76.47 | 73.94
  Weeks 9 to 10 | 83.30 | 82.20 | 83.82 | 76.11
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; This analysis refers to the test of the null hypothesis that there is no difference in the survival distribution function between the treatment groups; Test type: Superiority or Other; p = 0.1143, Generalized Wilcoxon
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.4544, Generalized Wilcoxon

2. Secondary Outcome: Change From Baseline in the Total HAM-A Score After 1 Week
Description: The Hamilton Anxiety (HAM-A) Rating scale is a test of 14 items measuring the severity of anxiety symptoms. Each item is rated on a 5-point ordinal scale, ranging from 0 (not present) to 4 (severe). Maximum HAM-A Score is 56.
Time Frame: Baseline and 1 week
Population: ITT population, but only subjects with values at baseline and time point are included in the analysis
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 112 | 109 | 63 | 57
Units on a scale | -9.3 (11.50) | -5.8 (9.04) | -7.8 (7.43) | -4.6 (8.33)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; ANCOVA with treatment as a fixed effect and baseline total HAM-A score as a covariate; Test type: Superiority or Other; p = 0.0173, ANCOVA
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; ANCOVA with treatment as a fixed effect and baseline total HAM-A score as a covariate; Test type: Superiority or Other; p = 0.0516, ANCOVA

3. Secondary Outcome: Change From Baseline in the Total HAM-A Score After 2 Weeks
Description: as for outcome 2
Time Frame: Baseline and 2 Weeks
Population: ITT Population, only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 108 | 103 | 61 | 53
Units on a scale | -11.6 (10.98) | -8.2 (9.37) | -10.0 (8.75) | -6.1 (9.06)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.0361, ANCOVA — P-value based on ANCOVA model with treatment as a fixed effect and baseline total HAM-A score as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.0366, ANCOVA — P-value based on ANCOVA model with treatment as a fixed effect and baseline total HAM-A score as a covariate

4. Secondary Outcome: Change From Baseline in the Total HAM-A Score After 3 Weeks
Description: as for outcome 2
Time Frame: Baseline and 3 weeks
Population: ITT population, only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 101 | 92 | 58 | 52
Units on a scale | -14.3 (11.81) | -12.9 (11.03) | -10.9 (9.70) | -9.5 (9.49)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.7390, ANCOVA — P-value based on ANCOVA model with treatment as a fixed effect and baseline total HAM-A score as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.6735, ANCOVA — P-value based on ANCOVA model with treatment as a fixed effect and baseline total HAM-A score as a covariate

5. Secondary Outcome: Change From Baseline in the Total HAM-A Score After 4 Weeks
Description: as for outcome 2
Time Frame: Baseline and 4 weeks
Population: ITT population, only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 97 | 90 | 54 | 48
Units on a scale | -15.2 (11.66) | -13.7 (10.58) | -12.9 (9.47) | -8.3 (8.35)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.4261, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline total HAM-A score as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.0231, ANCOVA — P-value based on ANCOVA with treatment as a fixed effect and baseline HAM-A score as a covariate

6. Secondary Outcome: Change From Baseline in the Total HAM-A Score After 5 Weeks
Description: as for outcome 2
Time Frame: Baseline and 5 weeks
Population: ITT population, only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 89 | 81 | 51 | 48
Units on a scale | -16.7 (11.81) | -14.4 (11.69) | -13.3 (8.41) | -10.3 (10.99)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.1820, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and total HAM-A score as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.2187, ANCOVA — P-value based on ANCOVA model with treatment as a fixed effect and baseline total HAM-A score as covariate

7. Secondary Outcome: Change From Baseline in the Total HAM-A Score After 6 Weeks
Description: as for outcome 2
Time Frame: Baseline and 6 weeks
Population: ITT population, only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 87 | 81 | 47 | 47
Units on a scale | -17.7 (11.94) | -15.1 (11.59) | -13.4 (8.00) | -11.0 (10.44)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.1456, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline total HAM-A score as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.3618, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline total HAM-A score as a covariate

8. Secondary Outcome: Change From Baseline in the Total HAM-A Score After 7 Weeks
Description: as for outcome 2
Time Frame: Baseline and 7 weeks
Population: ITT population, only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 83 | 82 | 53 | 49
Units on a scale | -17.7 (12.75) | -15.6 (11.78) | -13.3 (8.85) | -11.3 (11.32)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.3535, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline total HAM-A score as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.5660, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline total HAM-A score as a covariate

9. Secondary Outcome: Change From Baseline in the Total HAM-A Score After 8 Weeks
Description: as for outcome 2
Time Frame: Baseline and 8 weeks
Population: ITT population, only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 84 | 84 | 53 | 47
Units on a scale | -18.5 (13.38) | -16.6 (10.72) | -13.9 (8.71) | -12.3 (9.49)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.3414, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline total HAM-A score as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.7344, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline total HAM-A score as a covariate

10. Secondary Outcome: Change From Baseline in the Total HAM-A Score at Endpoint During the 8 Week Treatment Period
Description: The Hamilton Anxiety (HAM-A) Rating scale is a test of 14 items measuring the severity of anxiety symptoms. Each item is rated on a 5-point ordinal scale, ranging from 0 (not present) to 4 (severe). Maximum HAM-A Score is 56. Endpoint is last observed value during the 8 week treatment period.
Time Frame: Baseline and at endpoint during the 8 week treatment period
Population: ITT population, Last Observation Carried Forward imputation was applied
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 117 | 117 | 64 | 59
Units on a scale | -17.3 (13.03) | -14.3 (11.32) | -13.6 (8.85) | -11.5 (10.44)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.1197, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline total HAM-A score as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.4416, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline total HAM-A score as a covariate

11. Secondary Outcome: Clinical Response (Decrease From Baseline in Total HAM-A-score >=50%) After 1 Week
Description: The Hamilton Anxiety (HAM-A) Rating scale is a test of 14 items measuring the severity of anxiety symptoms. Each item is rated on a 5-point ordinal scale, ranging from 0 (not present) to 4 (severe).
Time Frame: 1 week
Population: ITT population, but only patients with a non-missing value at timepoint are included in the analysis
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 112 | 109 | 63 | 57
participants
  Response | 39 | 24 | 22 | 16
  No Response | 73 | 85 | 41 | 41
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Analysis refers to test of differences in response rates; Test type: Superiority or Other; p = 0.0350, Chi-squared
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Analysis refers to test of differences in response rates; Test type: Superiority or Other; p = 0.4205, Chi-squared

12. Secondary Outcome: Clinical Response (Decrease From Baseline in Total HAM-A-score >=50%) After 2 Weeks
Description: as for outcome 11
Time Frame: 2 weeks
Population: ITT population, but only patients with a non-missing value at timepoint are included in the analysis
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 108 | 103 | 61 | 53
participants
  Response | 48 | 38 | 30 | 23
  No Response | 60 | 65 | 31 | 30
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Analysis refers to test of differences in response rates; Test type: Superiority or Other; p = 0.2645, Chi-squared
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Analysis refers to test of differences in response rates; Test type: Superiority or Other; p = 0.5369, Chi-squared

13. Secondary Outcome: Clinical Response (Decrease From Baseline in Total HAM-A-score >=50%) After 3 Weeks
Description: as for outcome 11
Time Frame: 3 weeks
Population: ITT population, but only patients with a non-missing value at timepoint are included in the analysis
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 101 | 92 | 58 | 52
participants
  Response | 56 | 51 | 33 | 31
  No Response | 45 | 41 | 25 | 21
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Analysis refers to test of differences in response rates; Test type: Superiority or Other; p = 0.9988, Chi-squared
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Analysis refers to test of differences in response rates; Test type: Superiority or Other; p = 0.7729, Chi-squared

14. Secondary Outcome: Clinical Response (Decrease From Baseline in Total HAM-A-score >=50%) After 4 Weeks
Description: as for outcome 11
Time Frame: 4 weeks
Population: ITT population, but only patients with a non-missing value at timepoint are included in the analysis
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 97 | 90 | 54 | 48
participants
  Response | 58 | 56 | 37 | 25
  No Response | 39 | 34 | 17 | 23
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Analysis refers to test of differences in response rates; Test type: Superiority or Other; p = 0.7338, Chi-squared
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Analysis refers to test of differences in response rates; Test type: Superiority or Other; p = 0.0897, Chi-squared

15. Secondary Outcome: Clinical Response (Decrease From Baseline in Total HAM-A-score >=50%) After 5 Weeks
Description: as for outcome 11
Time Frame: 5 weeks
Population: ITT population, but only patients with a non-missing value at timepoint are included in the analysis
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 89 | 81 | 51 | 48
participants
  Response | 59 | 51 | 33 | 30
  Non Response | 30 | 30 | 18 | 18
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Analysis refers to test of differences in response rates; Test type: Superiority or Other; p = 0.6501, Chi-squared
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Analysis refers to test of differences in response rates; Test type: Superiority or Other; p = 0.8196, Chi-squared

16. Secondary Outcome: Clinical Response (Decrease From Baseline in Total HAM-A-score >=50%) After 6 Weeks
Description: as for outcome 11
Time Frame: 6 weeks
Population: ITT population, but only patients with a non-missing value at timepoint are included in the analysis
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 87 | 81 | 47 | 47
participants
  Response | 63 | 56 | 31 | 32
  No Response | 24 | 25 | 16 | 15
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Analysis refers to test of differences in response rates; Test type: Superiority or Other; p = 0.6404, Chi-squared
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Analysis refers to test of differences in response rates; Test type: Superiority or Other; p = 0.8263, Chi-squared

17. Secondary Outcome: Clinical Response (Decrease From Baseline in Total HAM-A-score >=50%) After 7 Weeks
Description: as for outcome 11
Time Frame: 7 weeks
Population: ITT population, but only patients with a non-missing value at timepoint are included in the analysis
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 83 | 82 | 53 | 49
participants
  Response | 60 | 57 | 37 | 34
  No Response | 23 | 25 | 16 | 15
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Analysis refers to test of differences in response rates; Test type: Superiority or Other; p = 0.6946, Chi-squared
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Analysis refers to test of differences in response rates; Test type: Superiority or Other; p = 0.9629, Chi-squared

18. Secondary Outcome: Clinical Response (Decrease From Baseline in Total HAM-A-score >=50%) After 8 Weeks
Description: as for outcome 11
Time Frame: 8 weeks
Population: ITT population, but only patients with a non-missing value at timepoint are included in the analysis
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 84 | 84 | 53 | 47
participants
  Response | 61 | 62 | 38 | 35
  No Response | 23 | 22 | 15 | 12
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Analysis refers to test of differences in response rates; Test type: Superiority or Other; p = 0.8617, Chi-squared
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Analysis refers to test of differences in response rates; Test type: Superiority or Other; p = 0.7555, Chi-squared

19. Secondary Outcome: Clinical Response (Decrease From Baseline in Total HAM-A-score >=50%) at Endpoint During the 8 Week Treatment Period
Description: The Hamilton Anxiety (HAM-A) Rating scale is a test of 14 items measuring the severity of anxiety symptoms. Each item is rated on a 5-point ordinal scale, ranging from 0 (not present) to 4 (severe). Endpoint is last observed value during the 8 week treatment period.
Time Frame: at endpoint during the 8 week treatment period
Population: ITT population, Last Observation Carried Forward imputation was applied
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 117 | 117 | 64 | 59
participants
  Response | 78 | 74 | 44 | 40
  No Response | 39 | 43 | 20 | 19
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Analysis refers to test of differences in response rates; Test type: Superiority or Other; p = 0.5836, Chi-squared
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Analysis refers to test of differences in response rates; Test type: Superiority or Other; p = 0.9096, Chi-squared

20. Secondary Outcome: Change in Severity of Illness From Baseline Using the Clinical Global Impression Improvement (CGI-I) Score After 2 Weeks
Description: The Clinical Global Impression Improvement (CGI-I) scale is a 7 point ordinal scale that assesses how the patient's illness has improved ranging from 'very much improved' to 'very much worse'(see definition of categories in results table).
Time Frame: Baseline and 2 weeks
Population: ITT population, but only patients with non-missing values were included
Measure: Number; unit: Participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 119 | 107 | 66 | 57
Participants
  Very much improved | 6 | 1 | 4 | 2
  much improved | 38 | 23 | 25 | 10
  minimally improved | 53 | 35 | 27 | 20
  No change | 17 | 40 | 9 | 18
  Minimally worse | 4 | 7 | 1 | 6
  Much worse | 1 | 1 | 0 | 1
  Very much worse | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; van Elteren test stratified by CGI-Severity score at baseline and testing between treatment differences in percentages based on non-missing responses within a timepoint. CGI-Severity score categorizes severity at baseline as normal,not at all ill, borderline mentally ill, mildly ill, moderately ill, markedly ill, severely ill, among the most extremely ill; Test type: Superiority or Other; p = 0.0002, van Elteren test
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.0006, van Elteren test

21. Secondary Outcome: Change in Severity of Illness From Baseline Using the Clinical Global Impression - Improvement (CGI-I) Score After 4 Weeks
Description: as for outcome 20
Time Frame: Baseline and 4 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 107 | 99 | 60 | 46
participants
  Very much improved | 18 | 5 | 12 | 1
  Much improved | 40 | 40 | 26 | 18
  Minimally improved | 35 | 23 | 13 | 17
  No change | 7 | 19 | 7 | 9
  Minimally worse | 6 | 9 | 1 | 1
  Much worse | 1 | 2 | 0 | 0
  Very much worse | 0 | 1 | 1 | 0
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; van Elteren test stratified by CGI-Severity score at baseline and testing between treatment differences in percentages based on non-missing responses within a timepoint, CGI-Severity score categorizes severity at baseline as normal,not at all ill, borderline mentally ill, mildly ill, moderately ill, markedly ill, severely ill, among the most extremely ill; Test type: Superiority or Other; p = 0.0255, van Elteren test
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.0065, van Elteren test

22. Secondary Outcome: Change in Severity of Illness From Baseline Using the Clinical Global Impression - Improvement (CGI-I) Score After 8 Weeks
Description: as for outcome 20
Time Frame: Baseline and 8 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 93 | 96 | 57 | 51
participants
  Very much improved | 28 | 27 | 14 | 12
  Much improved | 44 | 27 | 25 | 22
  Minimally improved | 16 | 19 | 11 | 13
  No change | 3 | 19 | 5 | 4
  Minimally worse | 2 | 1 | 1 | 0
  Much worse | 0 | 2 | 1 | 0
  Very much worse | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; van Elteren test stratified by CGI-Severity score at baseline and testing between treatment differences in percentages on non-missing responses within a timepoint. CGI-Severity score categorizes severity at baseline as normal,not at all ill, borderline mentally ill, mildly ill, moderately ill, markedly ill, severely ill, among the most extremely ill; Test type: Superiority or Other; p = 0.0370, van Elteren test
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.9569, van Elteren test

23. Secondary Outcome: Change in Severity of Illness From Baseline Using the Clinical Global Impression - Improvement (CGI-I) Score at Endpoint During the 8 Week Treatment Period
Description: The Clinical Global Impression Improvement (CGI-I) scale is a 7 point ordinal scale that assesses how the patient's illness has improved ranging from 'very much improved' to 'very much worse'(see definition of categories in results table). Endpoint is last observed value during the 8 week treatment period.
Time Frame: Baseline and at endpoint during the 8 week treatment period
Population: ITT population, but only subjects with non-missing values have been included
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 122 | 113 | 66 | 59
participants
  Very much improved | 31 | 27 | 14 | 12
  Much improved | 47 | 31 | 29 | 23
  Minimally improved | 30 | 24 | 12 | 16
  No change | 7 | 25 | 8 | 5
  Minimally worse | 6 | 2 | 2 | 2
  Much worse | 1 | 3 | 1 | 1
  Very much worse | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.0978, van Elteren test
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.7096, van Elteren test

24. Secondary Outcome: Subject's Assessment of Treatment Effect as Measured by the Patient Global Impression (PGI) Score After 1 Week
Description: The Patient Global Impression (PGI) scale is a 7 point ordinal scale that rates subject's assessment of treatment effect ranging from 'very much better' to 'very much worse' (see categories in results tables).
Time Frame: 1 week
Population: ITT population, but only patients with non-missing values are included in the analysis
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 109 | 102 | 61 | 53
participants
  Very much better | 7 | 0 | 3 | 0
  Much better | 24 | 5 | 10 | 7
  A little better | 35 | 40 | 27 | 9
  Unchanged | 39 | 46 | 20 | 31
  A little worse | 2 | 6 | 1 | 3
  Much worse | 1 | 5 | 0 | 2
  Very much worse | 1 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.0001, van Elteren test
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.0003, van Elteren test

25. Secondary Outcome: Subject's Assessment of Treatment Effect as Measured by the Patient Global Impression (PGI) Score After 2 Weeks
Description: The Patient Global Impression (PGI) scale is a 7 point ordinal scale that rates subject's assessment of treatment effect.
Time Frame: 2 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 110 | 104 | 62 | 54
participants
  Very much better | 10 | 2 | 5 | 4
  Much better | 30 | 16 | 21 | 7
  A little better | 34 | 38 | 21 | 20
  Unchanged | 29 | 37 | 13 | 17
  A little worse | 3 | 3 | 0 | 3
  Much worse | 4 | 5 | 1 | 2
  Very much worse | 0 | 3 | 1 | 1
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.0025, van Elteren test
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.0101, van Elteren test

26. Secondary Outcome: Subject's Assessment of Treatment Effect as Measured by the Patient Global Impression (PGI) Score After 3 Weeks
Description: as for outcome 24
Time Frame: 3 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 107 | 95 | 61 | 53
participants
  Very much better | 22 | 7 | 10 | 2
  Much better | 23 | 21 | 21 | 14
  A little better | 33 | 28 | 16 | 22
  Unchanged | 24 | 31 | 12 | 13
  A little worse | 2 | 3 | 1 | 0
  Much worse | 1 | 5 | 1 | 1
  Very much worse | 2 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.0095, van Elteren test
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.0390, van Elteren test

27. Secondary Outcome: Subject's Assessment of Treatment Effect as Measured by the Patient Global Impression (PGI) Score After 4 Weeks
Description: as for outcome 24
Time Frame: 4 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 102 | 93 | 57 | 49
participants
  Very much better | 18 | 13 | 13 | 6
  Much better | 38 | 24 | 19 | 14
  A little better | 26 | 20 | 16 | 18
  Unchanged | 14 | 28 | 5 | 8
  A little worse | 2 | 4 | 2 | 1
  Much worse | 2 | 3 | 2 | 1
  Very much worse | 2 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.0160, van Elteren test
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.1024, van Elteren test

28. Secondary Outcome: Subject's Assessment of Treatment Effect as Measured by the Patient Global Impression (PGI) Score After 5 Weeks
Description: as for outcome 24
Time Frame: 5 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 94 | 84 | 54 | 49
participants
  Very much better | 21 | 10 | 13 | 5
  Much better | 32 | 27 | 19 | 20
  A little better | 16 | 19 | 18 | 10
  Unchanged | 16 | 19 | 4 | 12
  A little worse | 3 | 2 | 0 | 1
  Much worse | 6 | 6 | 0 | 0
  Very much worse | 0 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.0761, van Elteren test
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.0376, van Elteren test

29. Secondary Outcome: Subject's Assessment of Treatment Effect as Measured by the Patient Global Impression (PGI) Score After 6 Weeks
Description: as for outcome 24
Time Frame: 6 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 93 | 84 | 50 | 48
participants
  Very much better | 22 | 16 | 15 | 6
  Much better | 29 | 24 | 20 | 15
  A little better | 23 | 17 | 11 | 16
  Unchanged | 16 | 18 | 4 | 8
  A little worse | 2 | 2 | 0 | 2
  Much worse | 1 | 5 | 0 | 0
  Very much worse | 0 | 2 | 0 | 1
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.1196, van Elteren test
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; van Elteren test stratified by CGI-Severity score at baseline and testing between treatment differences in percentages based on non-missing responses within a timepoint.CGI-Severity score categorizes severity at baseline as normal,not at all ill, borderline mentally ill, mildly ill, moderately ill, markedly ill, severely ill, among the most extremely ill; Test type: Superiority or Other; p = 0.0029, van Elteren test

30. Secondary Outcome: Subject's Assessment of Treatment Effect as Measured by the Patient Global Impression (PGI) Score After 7 Weeks
Description: as for outcome 24
Time Frame: 7 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 88 | 84 | 56 | 50
participants
  Very much better | 23 | 21 | 12 | 8
  Much better | 28 | 24 | 23 | 23
  A little better | 17 | 17 | 11 | 7
  Unchanged | 15 | 18 | 8 | 9
  A little worse | 3 | 1 | 2 | 1
  Much worse | 2 | 1 | 0 | 1
  Very much worse | 0 | 2 | 0 | 1
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.6323, van Elteren test
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.5533, van Elteren test

31. Secondary Outcome: Subject's Assessment of Treatment Effect as Measured by the Patient Global Impression (PGI) Score After 8 Weeks
Description: as for outcome 24
Time Frame: 8 weeks
Population: ITT population, Last Observation Carried Forward imputation was applied
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 88 | 86 | 56 | 48
participants
  Very much better | 28 | 23 | 20 | 13
  Much better | 28 | 22 | 14 | 13
  A little better | 17 | 21 | 13 | 12
  Unchanged | 13 | 16 | 8 | 7
  A little worse | 2 | 0 | 1 | 1
  Much worse | 0 | 3 | 0 | 1
  Very much worse | 0 | 1 | 0 | 1
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.1705, van Elteren test
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.3196, van Elteren test

32. Secondary Outcome: Subject's Assessment of Treatment Effect as Measured by the Patient Global Impression (PGI) Score at Endpoint During the 8 Week Treatment Period
Description: The Patient Global Impression (PGI) scale is a 7 point ordinal scale that rates subject's assessment of treatment effect ranging from 'very much better' to 'very much worse' (see categories in results tables). Endpoint is last observed value during the 8 week treatment period.
Time Frame: at endpoint during the 8 week treatment period
Population: ITT population, Last Observation Carried Forward imputation was applied
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 123 | 119 | 66 | 60
participants
  Very much better | 34 | 25 | 21 | 14
  Much better | 36 | 27 | 14 | 15
  A little better | 27 | 30 | 17 | 14
  Unchanged | 20 | 30 | 12 | 11
  A little worse | 3 | 0 | 1 | 1
  Much worse | 3 | 6 | 1 | 3
  Very much worse | 0 | 1 | 0 | 2
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.0419, van Elteren test
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.2541, van Elteren test

33. Secondary Outcome: Change From Baseline in HAM-A-insomnia Subscore After 1 Week
Description: The Hamilton Anxiety (HAM-A) Rating scale is a test of 14 items measuring the severity of anxiety symptoms. Each item is rated on a 5-point ordinal scale, ranging from 0 (not present) to 4 (severe). Maximum score of the insomnia subscore is 4.
Time Frame: Baseline and 1 week
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 112 | 109 | 63 | 57
Units on a scale | -0.9 (1.42) | -0.6 (1.43) | -1.0 (1.40) | -0.5 (1.40)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.0677, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAM-A insomnia subscore as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.0273, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAM-A insomnia subscore as a covariate

34. Secondary Outcome: Change From Baseline in HAM-A-insomnia Subscore After 2 Weeks
Description: as for outcome 33
Time Frame: Baseline and 2 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 108 | 103 | 61 | 53
Units on a scale | -1.0 (1.49) | -0.9 (1.40) | -1.2 (1.50) | -0.6 (1.50)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.5153, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAM-A insomnia subscore as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.0122, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAM-A insomnia subscore as a covariate

35. Secondary Outcome: Change From Baseline in HAM-A-insomnia Subscore After 3 Weeks
Description: as for outcome 33
Time Frame: Baseline and 3 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 101 | 92 | 58 | 52
Units on a scale | -1.2 (1.48) | -1.1 (1.43) | -1.4 (1.40) | -1.2 (1.36)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.4648, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAM-A insomnia subscore as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.5502, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAM-A insomnia subscore as a covariate

36. Secondary Outcome: Change From Baseline in HAM-A-insomnia Subscore After 4 Weeks
Description: as for outcome 33
Time Frame: Baseline and 4 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 97 | 90 | 54 | 48
Units on a scale | -1.3 (1.65) | -1.4 (1.47) | -1.6 (1.34) | -1.1 (1.42)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.9093, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAM-A insomnia subscore as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.1354, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAM-A insomnia subscore as a covariate

37. Secondary Outcome: Change From Baseline in HAM-A-insomnia Subscore After 5 Weeks
Description: as for outcome 33
Time Frame: Baseline and 5 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 89 | 81 | 51 | 48
Units on a scale | -1.3 (1.56) | -1.4 (1.52) | -1.5 (1.36) | -1.1 (1.22)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.7434, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAM-A insomnia subscore as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.1148, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAM-A insomnia subscore as a covariate

38. Secondary Outcome: Change From Baseline in HAM-A-insomnia Subscore After 6 Weeks
Description: as for outcome 33
Time Frame: Baseline and 6 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 87 | 81 | 47 | 47
Units on a scale | -1.4 (1.64) | -1.5 (1.52) | -1.6 (1.25) | -1.1 (1.39)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.9346, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAMA-A insomnia subscore as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.2709, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAM-A insomnia subscore as a covariate

39. Secondary Outcome: Change From Baseline in HAM-A-insomnia Subscore After 7 Weeks
Description: as for outcome 33
Time Frame: Baseline and 7 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 83 | 82 | 53 | 49
Units on a scale | -1.5 (1.63) | -1.4 (1.49) | -1.6 (1.32) | -1.2 (1.40)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.3827, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAM-A insomnia subscore as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.2513, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAM-A insomnia subscore as a covariate

40. Secondary Outcome: Change From Baseline in HAM-A-insomnia Subscore After 8 Weeks
Description: as for outcome 33
Time Frame: Baseline and 8 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 84 | 84 | 53 | 47
Units on a scale | -1.6 (1.57) | -1.6 (1.41) | -1.6 (1.33) | -1.3 (1.41)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.3930, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAM-A insomnia subscore as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.5461, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAM-A insomnia subscore as a covariate

41. Secondary Outcome: Change From Baseline in HAM-A-insomnia Subscore at Endpoint During the 8 Week Treatment Period
Description: The Hamilton Anxiety (HAM-A) Rating scale is a test of 14 items measuring the severity of anxiety symptoms. Each item is rated on a 5-point ordinal scale, ranging from 0 (not present) to 4 (severe). Maximum score of the insomnia subscore is 4. Endpoint is last observed value during the 8 week treatment period.
Time Frame: Baseline and at endpoint during the 8 week treatment period
Population: ITT population, Last Observation Carried Forward imputation was applied
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 117 | 117 | 64 | 59
Units on a scale | -1.6 (1.53) | -1.4 (1.49) | -1.5 (1.38) | -1.3 (1.51)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.0722, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAM-A insomnia subscore as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.4639, ANCOVA — P-values based on an ANCOVA with treatment as a fixed effect and baseline HAM-A insomnia subscore as a covariate

42. Secondary Outcome: Change From Baseline in HAM-A-psychic Factors Subscore After 1 Week
Description: The Hamilton Anxiety (HAM-A) Rating scale is a test of 14 items measuring the severity of anxiety symptoms. Each item is rated on a 5-point ordinal scale, ranging from 0 (not present) to 4 (severe). Maximum score of the psychic factors subscore is 4.
Time Frame: Baseline and 1 week
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 112 | 109 | 63 | 57
Units on a scale | -4.9 (5.73) | -2.9 (4.78) | -4.5 (4.53) | -3.3 (4.08)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.0075, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAMA-A psychic factors subscore as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.1641, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAM-A psychic factors subscore as a covariate

43. Secondary Outcome: Change From Baseline in HAM-A-psychic Factors Subscore After 2 Weeks
Description: as for outcome 42
Time Frame: Baseline and 2 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 108 | 103 | 61 | 53
Units on a scale | -6.0 (5.97) | -4.5 (4.88) | -5.8 (5.23) | -4.1 (4.53)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.0932, ANCOVA — [p-value comment as in outcome 42, analysis 1]
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.0852, ANCOVA — [p-value comment as in outcome 42, analysis 1]

44. Secondary Outcome: Change From Baseline in HAM-A-psychic Factors Subscore After 3 Weeks
Description: as for outcome 42
Time Frame: Baseline and 3 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 101 | 92 | 58 | 52
Units on a scale | -7.3 (5.98) | -6.8 (5.42) | -6.4 (5.44) | -6.1 (4.87)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.7896, ANCOVA — [p-value comment as in outcome 42, analysis 1]
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.9651, ANCOVA — [p-value comment as in outcome 42, analysis 1]

45. Secondary Outcome: Change From Baseline in HAM-A-psychic Factors Subscore After 4 Weeks
Description: as for outcome 42
Time Frame: Baseline and 4 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 97 | 90 | 54 | 48
Units on a scale | -7.7 (5.95) | -7.4 (5.57) | -7.8 (5.14) | -5.9 (4.80)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.8280, ANCOVA — [p-value comment as in outcome 42, analysis 1]
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.0936, ANCOVA — [p-value comment as in outcome 42, analysis 1]

46. Secondary Outcome: Change From Baseline in HAM-A-psychic Factors Subscore After 5 Weeks
Description: as for outcome 42
Time Frame: Baseline and 5 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 89 | 81 | 51 | 48
Units on a scale | -8.7 (5.84) | -7.7 (5.99) | -7.9 (5.08) | -6.8 (5.76)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.3539, ANCOVA — [p-value comment as in outcome 42, analysis 1]
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.4672, ANCOVA — [p-value comment as in outcome 42, analysis 1]

47. Secondary Outcome: Change From Baseline in HAM-A-psychic Factors Subscore After 6 Weeks
Description: as for outcome 42
Time Frame: Baseline and 6 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 87 | 81 | 47 | 47
Units on a scale | -9.4 (5.84) | -8.3 (5.66) | -8.7 (4.81) | -7.2 (5.82)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.2550, ANCOVA — [p-value comment as in outcome 42, analysis 1]
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.3125, ANCOVA — [p-value comment as in outcome 42, analysis 1]

48. Secondary Outcome: Change From Baseline in HAM-A-psychic Factors Subscore After 7 Weeks
Description: as for outcome 42
Time Frame: Baseline and 7 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 83 | 82 | 53 | 49
Units on a scale | -9.6 (6.27) | -8.4 (5.75) | -8.1 (5.16) | -7.6 (6.19)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.3174, ANCOVA — [p-value comment as in outcome 42, analysis 1]
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.9427, ANCOVA — [p-value comment as in outcome 42, analysis 1]

49. Secondary Outcome: Change From Baseline in HAM-A-psychic Factors Subscore After 8 Weeks
Description: as for outcome 42
Time Frame: Baseline and 8 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 84 | 84 | 53 | 47
Units on a scale | -9.9 (6.63) | -8.9 (5.13) | -8.5 (4.91) | -8.5 (5.51)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.3252, ANCOVA — [p-value comment as in outcome 42, analysis 1]
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.6090, ANCOVA — [p-value comment as in outcome 42, analysis 1]

50. Secondary Outcome: Change From Baseline in HAM-A-psychic Factors Subscore at Endpoint During the 8 Week Treatment Period
Description: The Hamilton Anxiety (HAM-A) Rating scale is a test of 14 items measuring the severity of anxiety symptoms. Each item is rated on a 5-point ordinal scale, ranging from 0 (not present) to 4 (severe). Maximum score of the psychic factors subscore is 4. Endpoint is last observed value during the 8 week treatment period.
Time Frame: Baseline and at endpoint during the 8 week treatment period
Population: ITT population, Last Observation Carried Forward imputation was applied
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 117 | 117 | 64 | 59
Units on a scale | -9.1 (6.58) | -7.6 (5.82) | -7.9 (5.19) | -7.9 (5.81)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.1247, ANCOVA — [p-value comment as in outcome 42, analysis 1]
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.8430, ANCOVA — [p-value comment as in outcome 42, analysis 1]

51. Secondary Outcome: Change From Baseline in HAM-A-somatic Subscore After 1 Week
Description: The Hamilton Anxiety (HAM-A) Rating scale is a test of 14 items measuring the severity of anxiety symptoms. Each item is rated on a 5-point ordinal scale, ranging from 0 (not present) to 4 (severe). Maximum score of the somatic subscore is 4.
Time Frame: Baseline and 1 week
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 112 | 109 | 63 | 57
Units on a scale | -4.4 (6.95) | -2.9 (5.80) | -3.3 (4.46) | -1.4 (5.43)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.1031, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAMA-A somatic subscore as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.0543, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAMA-A somatic subscore as a covariate

52. Secondary Outcome: Change From Baseline in HAM-A-somatic Subscore After 2 Weeks
Description: as for outcome 51
Time Frame: Baseline and 2 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 108 | 103 | 61 | 53
Units on a scale | -5.6 (6.31) | -3.7 (6.18) | -4.2 (5.52) | -2.0 (6.05)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.0508, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAMA-A somatic subscore as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.0871, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAMA-A somatic subscore as a covariate

53. Secondary Outcome: Change From Baseline in HAM-A-somatic Subscore After 3 Weeks
Description: as for outcome 51
Time Frame: Baseline and 3 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 101 | 92 | 58 | 52
Units on a scale | -7.0 (7.03) | -6.1 (7.55) | -4.5 (5.85) | -3.4 (6.27)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.8318, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAMA-A somatic subscore as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.5375, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAMA-A somatic subscore as a covariate

54. Secondary Outcome: Change From Baseline in HAM-A-somatic Subscore After 4 Weeks
Description: as for outcome 51
Time Frame: Baseline and 4 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 97 | 90 | 54 | 48
Units on a scale | -7.5 (6.96) | -6.4 (6.50) | -5.1 (5.95) | -2.3 (5.71)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.2186, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAMA-A somatic subscore as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.0422, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAMA-A somatic subscore as a covariate

55. Secondary Outcome: Change From Baseline in HAM-A-somatic Subscore After 5 Weeks
Description: as for outcome 51
Time Frame: Baseline and 5 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 89 | 81 | 51 | 48
Units on a scale | -8.0 (7.21) | -6.8 (7.14) | -5.4 (5.31) | -3.4 (6.95)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.1164, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAMA-A somatic subscore as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.1935, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAMA-A somatic subscore as a covariate

56. Secondary Outcome: Change From Baseline in HAM-A-somatic Subscore After 6 Weeks
Description: as for outcome 51
Time Frame: Baseline and 6 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 87 | 81 | 47 | 47
Units on a scale | -8.3 (7.41) | -6.8 (7.32) | -4.7 (4.83) | -3.8 (6.19)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.1244, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAMA-A somatic subscore as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.6182, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAMA-A somatic subscore as a covariate

57. Secondary Outcome: Change From Baseline in HAM-A-somatic Subscore After 7 Weeks
Description: as for outcome 51
Time Frame: Baseline and 7 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 83 | 82 | 53 | 49
Units on a scale | -8.1 (7.74) | 7.2 (7.38) | -5.2 (5.37) | -3.7 (6.64)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.4589, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAMA-A somatic subscore as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.3930, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAMA-A somatic subscore as a covariate

58. Secondary Outcome: Change From Baseline in HAM-A-somatic Subscore After 8 Weeks
Description: as for outcome 51
Time Frame: Baseline and 8 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 84 | 84 | 53 | 47
Units on a scale | -8.6 (7.98) | -7.7 (7.43) | -5.5 (5.53) | -3.8 (5.76)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.4450, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAMA-A somatic subscore as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.2924, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAMA-A somatic subscore as a covariate

59. Secondary Outcome: Change From Baseline in HAM-A-somatic Subscore at Endpoint During the 8 Week Treatment Period
Description: The Hamilton Anxiety (HAM-A) Rating scale is a test of 14 items measuring the severity of anxiety symptoms. Each item is rated on a 5-point ordinal scale, ranging from 0 (not present) to 4 (severe). Maximum score of the somatic subscore is 4. Endpoint is last observed value during the 8 week treatment period.
Time Frame: Baseline and at endpoint during the 8 week treatment period
Population: ITT population, Last Observation Carried Forward imputation was applied
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 117 | 117 | 64 | 59
Units on a scale | -8.2 (7.86) | -6.7 (7.18) | -5.6 (5.72) | -3.6 (6.24)
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.2184, ANCOVA — P-value based on an ANCOVA model with treatment as a fixed effect and baseline HAMA-A somatic subscore as a covariate
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.1281, ANCOVA — [p-value comment as in outcome 42, analysis 1]

60. Secondary Outcome: Presence of Any Panic Attack(s) (for Subjects With Panic Disorder Only) After 1 Week
Time Frame: 1 week
Population: ITT population, but only patients with non-missing assessments were included
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 118 | 112 | 0 | 0
participants
  Any panic attack | 76 | 69 |  |
  No panic attack | 42 | 43 |  |
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; test of difference in percentage of subjects reporting any panic attack; Test type: Superiority or Other; p = 0.6602, Chi-squared

61. Secondary Outcome: Presence of Any Panic Attack(s) (for Subjects With Panic Disorder Only) After 2 Weeks
Time Frame: 2 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 114 | 106 | 0 | 0
participants
  Any panic attack | 60 | 60 |  |
  No panic attack | 54 | 46 |  |
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; test of difference in percentage of subjects reporting any panic attack; Test type: Superiority or Other; p = 0.5544, Chi-squared

62. Secondary Outcome: Presence of Any Panic Attack(s) (for Subjects With Panic Disorder Only) After 3 Weeks
Time Frame: 3 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 107 | 95 | 0 | 0
participants
  Any panic attack | 41 | 37 |  |
  No panic attack | 66 | 58 |  |
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; test of difference in percentage of subjects reporting any panic attack; Test type: Superiority or Other; p = 0.9269, Chi-squared

63. Secondary Outcome: Presence of Any Panic Attack(s) (for Subjects With Panic Disorder Only) After 4 Weeks
Time Frame: 4 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 103 | 93 | 0 | 0
participants
  Any panic attack | 43 | 43 |  |
  No panic attack | 60 | 50 |  |
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; test of difference in percentage of subjects reporting any panic attack; Test type: Superiority or Other; p = 0.5271, Chi-squared

64. Secondary Outcome: Presence of Any Panic Attack(s) (for Subjects With Panic Disorder Only) After 5 Weeks
Time Frame: 5 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 95 | 84 | 0 | 0
participants
  Any panic attack | 35 | 40 |  |
  No panic attack | 60 | 44 |  |
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; test of difference in percentage of subjects reporting any panic attack; Test type: Superiority or Other; p = 0.1447, Chi-squared

65. Secondary Outcome: Presence of Any Panic Attack(s) (for Subjects With Panic Disorder Only) After 6 Weeks
Time Frame: 6 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 93 | 84 | 0 | 0
participants
  Any panic attack | 36 | 33 |  |
  No panic attack | 57 | 51 |  |
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; Test type: Superiority or Other; p = 0.9375, Chi-squared — P-value from a Chi-squared test

66. Secondary Outcome: Presence of Any Panic Attack(s) (for Subjects With Panic Disorder Only) After 7 Weeks
Time Frame: 7 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 88 | 85 | 0 | 0
participants
  Any panic attack | 32 | 31 |  |
  No panic attack | 56 | 54 |  |
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; test of difference in percentage of subjects reporting any panic attack; Test type: Superiority or Other; p = 0.9883, Chi-squared

67. Secondary Outcome: Presence of Any Panic Attack(s) (for Subjects With Panic Disorder Only) After 8 Weeks
Time Frame: 8 weeks
Population: ITT population, but only subjects with non-missing values have been included
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 88 | 87 | 0 | 0
participants
  Any panic attack | 26 | 32 |  |
  No panic attack | 62 | 55 |  |
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; test of difference in percentage of subjects reporting any panic attack; Test type: Superiority or Other; p = 0.3093, Chi-squared

68. Secondary Outcome: Presence of Any Panic Attack(s) (for Subjects With Panic Disorder Only) at Endpoint During the 8 Week Treatment Period
Description: Endpoint is last observed value during the 8 week treatment period.
Time Frame: at endpoint during the 8 week treatment period
Population: ITT population, Last Observation Carried Forward imputation was applied
Measure: Number; unit: participants
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 123 | 120 | 0 | 0
participants
  Any panic attack | 47 | 50 |  |
  No panic attack | 76 | 70 |  |
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; test of difference in percentage of subjects reporting any panic attack; Test type: Superiority or Other; p = 0.5824, Chi-squared

69. Primary Outcome: Cumulative Percent of Participants Showing a Response in the Symptoms of Anxiety (Decrease in Total Hamilton Anxiety (HAM-A) -Score of >=50%) in the Per Protocol Population (Kaplan-Meier-estimates)
Description: The Hamilton Anxiety (HAM-A) Rating scale is a test of 14 items measuring the severity of anxiety symptoms. Each item is rated on a 5-point ordinal scale, ranging from 0 (not present) to 4 (severe). Total possible score is 56. Kaplan-Meier-analysis was performed and Kaplan-Meier estimates (cumulative percent of subjects responding) are presented.
Time Frame: 10 weeks
Population: Per Protocol Population (subjects of ITT population who have no major protocol violations)
Measure: Number; unit: cumulative percent of responders
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Number analyzed (Participants) | 104 | 106 | 53 | 49
cumulative percent of responders
  Week 1 | 1.92 | 0.94 | 1.89 | 2.04
  Week 2 | 35.58 | 24.53 | 33.96 | 30.78
  Week 3 | 51.23 | 41.54 | 52.83 | 53.16
  Week 4 | 63.18 | 54.19 | 58.49 | 67.21
  Week 5 | 75.45 | 67.59 | 67.92 | 71.89
  Week 6 | 77.59 | 71.94 | 71.70 | 79.56
  Week 7 | 79.83 | 75.77 | 77.70 | 79.56
  Week 8 | 80.95 | 78.32 | 79.93 | 79.56
  Week 9 to 10 | 86.60 | 84.82 | 86.62 | 82.48
Statistical Analysis 1: Comparison: Panic: Niravam+SSRI/SNRI vs Panic: SSRI/SNRI Alone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.044, Generalized Wilcoxon Test
Statistical Analysis 2: Comparison: GAD : Niravam+SSRI/SNRI vs GAD: SSRI/SNRI Alone; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.6587, Generalized Wilcoxon Test

ADVERSE EVENTS:
Description: The safety population consists of 414 subjects that received at least one dose of SSRI/SNRI and/or Niravam.
Arm/Group | Panic: Niravam+SSRI/SNRI | Panic: SSRI/SNRI Alone | GAD : Niravam+SSRI/SNRI | GAD: SSRI/SNRI Alone
Serious Adverse Events (participants affected / at risk) | 3/137 | 2/135 | 0/71 | 2/71
Other Adverse Events (participants affected / at risk) | 20/137 | 10/135 | 12/71 | 5/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Panic: Niravam+SSRI/SNRI (N=137) | Panic: SSRI/SNRI Alone (N=135) | GAD : Niravam+SSRI/SNRI (N=71) | GAD: SSRI/SNRI Alone (N=71)
Bronchitis acute (Infections and infestations) | 0 | 1 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0 | 0
Postoperative infection (Infections and infestations) | 1 | 0 | 0 | 0
Multiple drug overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Temporal Arteritis (Vascular disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Sternitis (Infections and infestations) | 1 | 0 | 0 | 0
Bacterial Pyelonephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panic: Niravam+SSRI/SNRI (N=137) | Panic: SSRI/SNRI Alone (N=135) | GAD : Niravam+SSRI/SNRI (N=71) | GAD: SSRI/SNRI Alone (N=71)
Headache (Nervous system disorders) | 8 | 5 | 4 | 4
Somnolence (Nervous system disorders) | 9 | 2 | 3 | 0
Fatigue (General disorders) | 3 | 3 | 5 | 1

LIMITATIONS AND CAVEATS:
Originally it was planned to enrol and randomize 848 subjects. The smaller than planned sample size was a result of an unusually high rate of screening failure (results published in Psychiatry 2006, Vol. 3, Issue 12 , pages 39 - 59).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.